CLINICAL TRIAL: NCT05032001
Title: ORAL ANTIDIABETICS EFFECT ON VISCERAL FAT MEASURED BY BIOIMPEDANCE IN TYPE 2 DIABETES PATIENTS. Pilot Study.
Brief Title: ORAL ANTIDIABETICS EFFECT ON VISCERAL FAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Metabolic Research Unit (Industry)
Responsible Party: Principal Investigator, Alonso Alberto Castro Arguelles, Metabolic Research Unit, Metabolic Research Unit
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: protocol1
Record Dates: First submitted 2021-08-21; First posted 2021-09-02 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity, Abdominal; Diabetes Mellitus, Type 2 | interventions — Biguanides; Dipeptidyl-Peptidase IV Inhibitors; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin (Experimental): Metformin 1.7-2.5mg per day during twelve weeks
  Interventions: Drug: Biguanide, DPP4 inhibitors, SGLT2 inhibitors
- Metformina + IDDP-4 (Experimental): Metformin 1.7-2.5mg per day plus Linagliptin 5mg per day or Sitagliptin 50-100mg per day
  Interventions: Drug: Biguanide, DPP4 inhibitors, SGLT2 inhibitors
- Metformina + ISGLT-2 (Experimental): Metformin 1.7-2.5mg per day plus Empaglifozin 10-25mg per day or Dapaglifozin 10mg per day
  Interventions: Drug: Biguanide, DPP4 inhibitors, SGLT2 inhibitors

INTERVENTIONS:
Drug: Biguanide, DPP4 inhibitors, SGLT2 inhibitors — Oral antidiabetic treatment during twelve weeks

SUMMARY:
Weight control is an essential part of treatment for type 2 diabetes (T2D) patients. Weight loss is associated with decreased haemoglobin A1c (A1c) levels. In particular, visceral fat is accompanied by more alterations in glucose and lipid metabolism. Quantification of visceral fat with bioimpedance (BIA) is closely related to measurement with computed axial tomography. Different available oral antidiabetics cause weight loss and total body fat (biguanides, DPP-4 inhibitors and SGLT-2 inhibitors), but it has only been shown that SLGT2 inhibitors decrease visceral fat. Therefore, the aim of this study is to determine whether there is a difference in the amount of visceral fat measured with BIA in T2D patients between three oral antidiabetic regimens after twelve weeks of treatment, to compare the effect on visceral fat between metformin, DPP4 inhibitors and SGLT2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients +18 years
* Patients with visceral fat quantification by BIA at baseline and week twelve
* Patients with body mass index >25
* Patients can swallow tablets

Exclusion Criteria:

* Patients treated with other oral antidiabetic agents or insulin
* Glomerular filtration rate less than 30 mL/min
* Transaminemia greater than 2 times the upper reference value
* Pregnancy
* Malnutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visceral fat measured by bioimpedance in kg at weet twelve | Baseline and week twelve
  Bioimpedance is a confident method to measured visceral fat

OTHER OUTCOMES:
Change from baseline in A1c level at week twelve | Baseline and week twelve
  Glycated hemoglobin percentage is the most reliable method to explain glycemic control in type 2 diabetes patients

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Research Unit, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee DH, Park KS, Ahn S, Ku EJ, Jung KY, Kim YJ, Kim KM, Moon JH, Choi SH, Park KS, Jang HC, Lim S. Comparison of Abdominal Visceral Adipose Tissue Area Measured by Computed Tomography with That Estimated by Bioelectrical Impedance Analysis Method in Korean Subjects. Nutrients. 2015 Dec 16;7(12):10513-24. doi: 10.3390/nu7125548. PMID 26694460
- [Background] Park KS, Lee DH, Lee J, Kim YJ, Jung KY, Kim KM, Kwak SH, Choi SH, Park KS, Jang HC, Lim S. Comparison between two methods of bioelectrical impedance analyses for accuracy in measuring abdominal visceral fat area. J Diabetes Complications. 2016 Mar;30(2):343-9. doi: 10.1016/j.jdiacomp.2015.10.014. Epub 2015 Oct 24. PMID 26620129
- [Background] Golay A. Metformin and body weight. Int J Obes (Lond). 2008 Jan;32(1):61-72. doi: 10.1038/sj.ijo.0803695. Epub 2007 Jul 24. PMID 17653063
- [Background] Nauck MA, Meininger G, Sheng D, Terranella L, Stein PP; Sitagliptin Study 024 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor, sitagliptin, compared with the sulfonylurea, glipizide, in patients with type 2 diabetes inadequately controlled on metformin alone: a randomized, double-blind, non-inferiority trial. Diabetes Obes Metab. 2007 Mar;9(2):194-205. doi: 10.1111/j.1463-1326.2006.00704.x. PMID 17300595
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392
- [Background] Sugiyama S, Jinnouchi H, Kurinami N, Hieshima K, Yoshida A, Jinnouchi K, Nishimura H, Suzuki T, Miyamoto F, Kajiwara K, Jinnouchi T. Dapagliflozin Reduces Fat Mass without Affecting Muscle Mass in Type 2 Diabetes. J Atheroscler Thromb. 2018 Jun 1;25(6):467-476. doi: 10.5551/jat.40873. Epub 2017 Dec 8. PMID 29225209
- [Background] Schork A, Saynisch J, Vosseler A, Jaghutriz BA, Heyne N, Peter A, Haring HU, Stefan N, Fritsche A, Artunc F. Effect of SGLT2 inhibitors on body composition, fluid status and renin-angiotensin-aldosterone system in type 2 diabetes: a prospective study using bioimpedance spectroscopy. Cardiovasc Diabetol. 2019 Apr 5;18(1):46. doi: 10.1186/s12933-019-0852-y. PMID 30953516
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476